CLINICAL TRIAL: NCT05989165
Title: Effectiveness of Combination Therapy of Microneedling and Minoxidil in Androgenetic Alopecia of Indonesian Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kara Adistri, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23030294
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Solutions; Percutaneous Collagen Induction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minoxidil 5% solution (Experimental): Patients will receive minoxidil 5%, twice a day, for a total duration of 12 weeks.
  Interventions: Drug: Minoxidil 5% Topical Solution
- Combination therapy of microneedling and minoxidil 5% solution (Experimental): Patients will receive a combination therapy of microneedling and minoxidil 5%. Minoxidil 5%, will be given twice a day for a total duration of 12 weeks. The microneedling treatment will be given every 4 weeks (week 0, week 4, week 8)for a total duration of 12 weeks.
  Interventions: Drug: Minoxidil 5% Topical Solution; Device: microneedling

INTERVENTIONS:
Drug: Minoxidil 5% Topical Solution — Patient will be given minoxidil 5% topical solution, twice a day for 12 weeks
Device: microneedling — Patient will be given microneedling treatment every 4 weeks
  Arms: Combination therapy of microneedling and minoxidil 5% solution

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of combination therapy of microneedling and minoxidil in androgenetic alopecia of Indonesian men. The main questions it aims to answer are:

* Is there an increase in hair density with combination therapy of microneedling and minoxidil versus minoxidil monotherapy?
* Is there an increase in hair diameter with combination therapy of microneedling and minoxidil versus minoxidil monotherapy?

Participants will be divided into 2 groups. The first one will receive minoxidil monotherapy, and the second one will receive a combination therapy of microneedling and minoxidil. Researchers will compare those 2 groups to see if there is a difference of effectiveness based on hair density and diameter.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Indonesian
* Age 18-59 years
* Diagnosis of androgenetic alopecia
* Hamilton-Norwood type III-IV

Exclusion Criteria:

* Use of minoxidil or finasteride topical 1 month prior
* Use of minoxidil or finasteride oral 1 month prior
* Skin infection in the treatment area
* Cosmetic procedures for the treatment of alopecia androgenetic such as platelet rich plasma, laser therapy,or microneedling 3 months prior
* History of keloid

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Density of hair | 12 weeks
  Increase density of hair in alopecia androgenetic patient
Diameter of hair | 12 weeks
  Increase diameter of hair in alopecia androgenetic patient

CONTACTS AND LOCATIONS:
Overall Officials: Kara Adistri, MD, Principal Investigator — Faculty of medicine, University of Indonesia
Locations (1):
- Cipto Mangungkusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dhurat R, Sukesh M, Avhad G, Dandale A, Pal A, Pund P. A randomized evaluator blinded study of effect of microneedling in androgenetic alopecia: a pilot study. Int J Trichology. 2013 Jan;5(1):6-11. doi: 10.4103/0974-7753.114700. PMID 23960389
- [Result] Kumar MK, Inamadar AC, Palit A. A Randomized Controlled, Single-Observer Blinded Study to Determine the Efficacy of Topical Minoxidil plus Microneedling versus Topical Minoxidil Alone in the Treatment of Androgenetic Alopecia. J Cutan Aesthet Surg. 2018 Oct-Dec;11(4):211-216. doi: 10.4103/JCAS.JCAS_130_17. PMID 30886475